CLINICAL TRIAL: NCT03136328
Title: Diagnosis and Staging of Neuroendocrine Tumors (NETs) Utilizing 68Ga-DOTATOC PET/CT Scan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: NCM USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-06-274
Record Dates: First submitted 2017-04-05; First posted 2017-05-02 (Actual); Results first posted 2019-01-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTATOC PET/CT (Experimental): Study participants will receive 68Ga-DOTATOC and undergo a PET/CT imaging study.
  Interventions: Drug: 68Ga-DOTATOC

INTERVENTIONS:
Drug: 68Ga-DOTATOC — The intervention is to administer 68Ga-DOTATOC PET/CT for detecting NET.
  Other Names: Diagnostic test

SUMMARY:
The primary goal of the analysis is to estimate the diagnostic accuracy of Gallium 68 (68Ga) -DOTATOC PET/CT for detecting neuroendocrine tumors (NETs) compared to conventional imaging techniques such as Magnetic Resonance Imaging (MRI) and Computerized Tomography (CT). Participants with histologically and/or clinically confirmed and/or suspected NET will be enrolled.

DETAILED DESCRIPTION:
This is a prospective, Phase 2, single center study of participants with Neuroendocrine Tumors (NETs). Study participants will receive 68Ga-DOTATOC. DOTATOC is a somatostatin analogue that localizes on the somatostatin receptors expressed by NETs and is attached to a radioactive material called Gallium 68. Participants will undergo a PET/CT imaging study to investigate 68Ga-DOTATOC's suitability as a positron emission tomography (PET) imaging agent for NETs. The radiation (imaging) dose will be 111-185 megabecquerel (MBq) (3 - 5 mCi) ± 25%. All doses after labeling will be presented in buffered solution for intravenous injection. Imaging will start 90 ±30 minutes after injection.

Sensitivity and specificity of this imaging technique will be compared with those of conventional imaging modality including CT, MRI and In-111 Octreoscan performed within 6-12 months before or after PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Patients of either gender, aged ≥18 years.
* Karnofsky status ≥60.
* Life expectancy of at least 12 weeks.
* Histologically and/or clinically confirmed and/or suspicious of NET.
* A diagnostic CT or MRI of the tumour region or suspected area within the previous 12 weeks prior to dosing day is available.
* Somatostatin-analogue scintigraphy scan with result (positive or negative) within the last 12 weeks.
* Recent Blood test results up to 4-6 weeks as follows:

  1. White Blood Cell (WBC): >2*109/L
  2. Haemoglobin: >8.0g/Dl
  3. Platelets: >50x109/L
  4. Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Alkaline phosphatase (AP) each less than, or equal to, 5 times its Upper Limit of Normal (ULN)
  5. Bilirubin less than, or equal to, three times its ULN
* Serum creatinine: within normal range or <120μmol/L for patients aged 60 years or older.
* Negative pregnancy test in women capable of child-bearing.

Exclusion Criteria:

* Known hypersensitivity to Gallium 68, DOTATOC or to any of the excipients of 68Ga-DOTATOC.
* Therapeutic use of any somatostatin analogue, including Sandostatin® LAR (Long Acting Release) (within 28 days) and Sandostatin® (within 2 days) prior to study imaging. If a patient is on Sandostatin® LAR a wash-out phase of 28 days is required before the injection of the study drug.
* Pregnant or breast-feeding women.
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charito Love, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Montefiore Medical Center which has medical specializing in the diagnosis and treatment of NETs. Eligible participants were those referred by their physicians for PET (Positron Emission Tomography) or CT imaging due to suspected or confirmed NETs.
Groups:
- 68Ga-DOTATOC PET/CT: Study participants will receive Gallium 68 (68Ga)-DOTATOC and undergo a PET/CT imaging study.
Period: Overall Study
Arm/Group | 68Ga-DOTATOC PET/CT
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 68Ga-DOTATOC PET/CT will be compared with final diagnoses for sensitivity, specificity and accuracy for detecting NET primary lesion and/or metastases. Results will be compared with conventional imaging results.
Groups:
- 68Ga-DOTATOC PET/CT: Study participants will receive 68Ga-DOTATOC and undergo a PET/CT imaging study to measure its ability to detect primary NET and any metastasis.
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity to Correctly Diagnose NET
Description: Sensitivity to detect NET will be assessed and compared with conventional imaging modality. Sensitivity is the ability of an agent to indicate the presence and location of NET. The ability of 68Ga-DOTATOC to localize more effectively to somatostatin receptors and the exquisite spatial resolution of PET/CT should make easier detection of primary and metastatic neuroendocrine tumors and allow better measurement of tumor burden. Sensitivity is the percentage of accurately diagnosed NET cases. All participants underwent conventional imaging with either Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) as standard care prior to 68Ga-DOTATOC imaging.
Time Frame: During imaging process ( approximately 120 minutes)
Measure: Number; unit: percent of NET correctly diagnosed
Groups:
- Conventional Imaging: All participants underwent conventional imaging with either Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) or In-111 Octreoscan as standard care prior to 68Ga-DOTATOC imaging.
Arm/Group | 68Ga-DOTATOC PET/CT | Conventional Imaging
Number analyzed (Participants) | 11 | 11
percent of NET correctly diagnosed
  Primary lesions | 75 | 75
  Liver metastases | 100 | 75
  Lymph node metastasis | 100 | 40
  Bone metastasis | 100 | 50

2. Secondary Outcome: Specificity to Detect True Negative
Description: A tumor is an abnormal growth of cells which can be malignant or not. NET tumors secrete hormones that will disrupt the normal ecology of the body. 68Ga-DOTATOC is extremely sensitive and specific to the receptors expressed by NET. These attributes are unique to 68Ga-DOTATOC and makes it the only imagining technique that can determine whether or not lesions detected by conventional imaging is due to NET involvement. 68Ga-DOTATOC is able to exclude disease involvement in lesions detected on CT/MRI; this ability to exclude disease involvement is called Specificity. The reported values indicate the specificity of 68Ga-DOTATOC, which is the percentage of tumors detected by conventional imagining that 68Ga-DOTATOC correctly determined were not due to NET involvement (i.e. identifying true negative for NET).
Time Frame: During imaging process ( approximately 120 minutes)
Measure: Number; unit: percent of tumors identified as non-NET
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 11
percent of tumors identified as non-NET
  Primary lesions | 100
  Liver metastases | 100

ADVERSE EVENTS:
Time Frame: The somatostatin analogue being administered is a short acting agent that, if it caused an adverse effect, would be seen within a few minutes after administration. Participants were monitored for one hour after injection. Participants were systematically assessed and questioned regarding changes in sensation or appearance of new symptom.
Arm/Group | 68Ga-DOTATOC PET/CT
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03136328/Prot_SAP_000.pdf